CLINICAL TRIAL: NCT00534014
Title: Vitamin C Therapy in Type 2 Diabetes and Cardiovascular Risk
Brief Title: Vitamin C and Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: David S. Schade, University of New Mexico
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 04-319B
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Atherosclerosis; Type 2 Diabetes
MeSH Terms: conditions — Atherosclerosis; Diabetes Mellitus, Type 2 | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Placebo Comparator): 0 mg of Vitamin C
  Interventions: Dietary Supplement: Vitamin C
- B (Active Comparator): 250 mg Vitamin C
  Interventions: Dietary Supplement: Vitamin C
- C (Active Comparator): 500 mg Vitamin C
  Interventions: Dietary Supplement: Vitamin C
- D (Active Comparator): 1000 mg Vitamin C
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Dietary Supplement: Vitamin C — Arm A = 0 mg Vitamin C, Arm B = 250 mg Vitamin C, Arm C = 500 mg Vitamin C, Arm D = 1000 mg Vitamin C

SUMMARY:
Study Goal #1: Determine the optimal oral dose of vitamin C to reduce surrogate markers of atherosclerosis (blockages in blood vessels) following the consumption of an atherogenic high fat lunch in type 2 diabetic individuals.

Study Goal #2: After conducting the original study, we found that vitamin E was not effective in reducing the markers of oxidative stress, hypercoagulation, inflammation, and metabolic parameters in patients with type 2 diabetes.

To date, data from randomized trials have largely demonstrated no significant benefit of vitamin E supplementation on the prevention of primary and/or secondary cardiovascular disease as once thought. Therefore, we decided to amend our current protocol to add a Part B to study only the effects of vitamin C at the following doses: 500 mg, 1000 mg, and 2000 mg daily (and include a placebo arm, as well.

DETAILED DESCRIPTION:
More than 70% of type 2 diabetic individuals will die of atherosclerotic disease (1). This is partially explained by the abnormal lipid profile frequently observed in type 2 diabetes. These patients are also frequently afflicted with "Syndrome X," an assortment of risk factors for atherosclerosis, including hypertension, abdominal obesity, hyperuricemia, prothrombotic and proinflammatory states, and increased plasminogen activator inhibitor type I (PAI-1) (2).

Several approaches have been suggested to reduce the risk of atherosclerosis in type 2 diabetic individuals. Changes in lifestyle leading to increased exercise and weight loss will result in the reduction of adipose stores (and restore tissue sensitivity to insulin). However, this approach is very difficult for many individuals to achieve. For them, this can be supplemented with medications such as aspirin, angiotensin inhibitors, angiotensin receptor blockers, and the statins. Unfortunately, each of these medications is either expensive and/or includes undesirable side effects (3). In addition, clinical experience shows that many patients are against taking medication for cultural reasons and/or fear of long-term unknown consequences.

For these reasons, there is great interest in using vitamins to reduce atherogenic risk. More than half of the U.S. adult population consumes vitamins on a regular basis. They are inexpensive and easily accessible in grocery stores and health food stores. The FDA does not consider them as "drugs" and they undergo a less rigorous approval procedure (4,5). Vitamins are natural compounds found in the body, and many individuals do not consider them drugs, but feel they are simply fortifying their bodies against disease.

There is currently a focus on vitamins that are antioxidants, including vitamin C. Patients with diabetes usually have a decreased antioxidant status, which leads to increased oxidative stress and vascular dysfunction (6,7). Oxidative stress refers to the excessive production of oxygen free radical species, which damage their surrounding molecules, and this leads to the increased release of inflammatory mediators, oxidation of low-density lipoproteins (LDL), and increased coagulation (7).

Vitamin C, another antioxidant, has been shown to regenerate Vitamin E, and in patients with increased oxidative stress (i.e. patients with conditions such as diabetes mellitus, coronary artery disease, and hypercholesterolemia), it restores endothelium-dependent artery vasodilation, and may reverse endothelial dysfunction in peripheral arteries (6). It has been hypothesized that supplementation of vitamin C may be more effective than vitamins taken together.

The hypothesis that atherosclerosis may be prevented by blocking the oxidative metabolism of LDL cholesterol, hence decreasing its uptake into the arterial lumen, is what incited the interest in vitamin C for treating coronary heart disease (CHD). Basic science and animal studies had shown beneficial effects of vitamin C on several different stages of the atherosclerotic process. This was followed by several observational studies on patients with no initial coronary artery disease, which suggested that vitamin C lowered the risk of future CHD. However, this was followed by several large randomized control trials, the majority of which showed no benefit of vitamin C in the prevention of CHD in patients with at least one coronary risk factor. However, this did not answer the question of whether vitamin C was beneficial in differeing doses.

In 2002, Fang et al. published a study that investigated the efficacy of vitamins C and E on the prevention of transplant-associated arteriosclerosis (another highly oxidative state). The primary outcome was change in average intimal index (plaque area divided by vessel area), which was measured with intavascular ultrasonography (IVUS). The vitamin C and E plasma concentrations were measured at baseline and at 1-year follow-up. At follow-up the placebo group showed a significant increase but the treatment group showed no change. The authors concluded that early progression of transplant-associated coronary arteriosclerosis is delayed with combined vitamin C and E therapy (6,10). In 2003, Salonen et al. published the six-year effects of combined vitamin C and E from the ASAP (Antioxidant Supplementation in Atherosclerosis Prevention) study, which studied the effects of supplemented doses on the progression of common carotid atherosclerosis in middle-aged high-risk men and women, using high-resolution ultrasound to assess this outcome. The group receiving combined vitamins showed a decrease in rate of progression of carotid intimal thickness, but this effect was limited to men only (8,10). In the Heart Protection Study (2002), a combination of synthetic vitamin E, vitamin C, and beta-carotene daily had no effect on the incidence of cardiovascular events in a group of approximately 20,000 high-risk individuals (10).

Therefore, not all studies showed positive benefits. Vitamin C has been shown to reduce overall oxidative stress by scavenging free readicals within the body (11). Some trials failed to report antioxidant levels, making compliance difficult to measure (8) (except through pill counting - and unfortunately, volunteers can dispose medications prior to visit, in order to give the image of compliance). Some trials used suboptimal timing regarding administration of antioxidant vitamins in relation to meals (1). Also, it is not known just what exactly is the optimal dosage of vitamins C is. The doses of vitamin C has differed in these trials (8); some investigators hypothesize that at least 500 mg/day of vitamin C are effective for slowing the progression of atherosclerosis, but speculation is rampant (7,8).

Based on the data from these studies (1,7,8), we believe that only sufficient doses of vitamins C will be effective for slowing the progression of atherosclerosis. It is our goal to find the optimal dosing combination. We will use a high-risk population (diabetic volunteers) because they are known to have high oxidative stress and may benefit tremendously from this therapy.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic for at lease 6 months
* Body mass index less than 40kg/m2
* Normal EEG's
* Normal test results from screening visit.

Exclusion Criteria:

* Known vascular disease
* Uncontrolled hypertension (>140/90 mmHg) or marked hyperlipidemia (serum low denisity lipoprotein >4.1 mmol/L or serum triglycerides > 7.8 mmol/L)
* Pregnancy
* Cigarette smoking
* Currently taking coumadin
* Recent use of antioxidant supplements or asprin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2007-03 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To determine the optimal oral dose of vitamin C and E to reduce surrogate markers of atherosclerosis (blockages in blood vessels) following the consumption of an atherogenic high fat lunch in type 2 diabetic individuals. | 8 weeks

SECONDARY OUTCOMES:
To study the effects of vitamin C on fibrinogen, insulin, glucose, PAI-1, adiponectin, free MDA, Oxy LDL,CRP, cholesterol, and FFA. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David S Schade, M.D., Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico , Clinical Translational Science Center, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Gutierrez AD, Duran-Valdez E, Robinson I, de Serna DG, Schade DS. Does short-term vitamin C reduce cardiovascular risk in type 2 diabetes? Endocr Pract. 2013 Sep-Oct;19(5):785-91. doi: 10.4158/EP12431.OR. PMID 23757614